CLINICAL TRIAL: NCT03063372
Title: Pomegranate Supplementation and Well-Being Among Medical Students and Residents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: University of Rhode Island (Other)
Responsible Party: Principal Investigator, Joshua Mann, Professor, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2016-0319
Record Dates: First submitted 2017-02-16; First posted 2017-02-24 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Antioxidant; Burnout, Professional; Psychological Distress
Keywords: Pomegranate; Burnout; Psychological Distress; Antioxidant
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Phase 1 is a single group feasibility pilot in 10 participants, all of whom will receive the nutritional supplement. Phase 2 is a parallel double blinded trial in 40 participants, half of whom will receive the supplement and half of whom will receive a placebo.
Who Masked: Participant, Investigator
Masking Description: Phase 1 is not masked, but in phase 2 the participants and investigator will be masked (double blind).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pomegranate Supplement (Experimental): Participants in this arm will take a capsule with 500 mg of "Pomella" pomegranate extract twice each day for 28 days.
  Interventions: Dietary Supplement: Pomella pomegranate extract
- Placebo (Placebo Comparator): Participants in this arm will take a gelatin placebo capsule twice each day for 28 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Pomella pomegranate extract — Participants will take a 500 mg capsule of pomegranate extract twice daily for 28 days.
  Arms: Pomegranate Supplement
Other: Placebo — Participants will take a gelatin placebo twice daily for 28 days.
  Arms: Placebo

SUMMARY:
Medical students and residents have high rates of mental distress and burnout related to the intellectual and time demands of their training. Research shows that physiological stress on the body can be a result of fatigue and high stress work, and is associated with experiences related to mental distress. Pomegranate is a fruit that is known to contain a variety of antioxidant substances that can reduce physiological stress. This study will look at the potential for pomegranate supplementation to reduce physiological stress and improve well-being in medical students and residents.

DETAILED DESCRIPTION:
This is a pilot study to investigate the feasibility of conducting a randomized trial of pomegranate supplementation in medical students and residents, and to see whether there is evidence of an effect on reported emotional and physical well-being.

Phase 1 will be a pilot with 10 participants in which all will receive the pomegranate supplement for 28 days. In phase 2, we will randomize 40 participants (1:1) to receive either the pomegranate supplement or a placebo.

For both phases, we will measure self reported emotional and physical well-being using several questionnaires, and we will conduct laboratory testing for measures of oxidative stress and inflammatory biomarkers in blood, and for a metabolite of pomegranate in urine.

ELIGIBILITY:
Inclusion Criteria:

* First or second year medical student or first or second year resident listed at the University of Mississippi Medical Center

Exclusion Criteria:

* Pregnant or planning to become pregnant during the study period.
* Breast feeding.
* Unable to speak, understand, and read English.
* Taking chronic medications other than contraception
* Taking supplements (including over-the-counter multivitamins)
* Allergy to pomegranate or gelatin (gel-caps)
* Baseline scores on the DASS-21 that indicate a level of depressive or anxiety symptoms that is "severe" or "extremely severe." This would be a depression score greater than 10, or an anxiety score greater than 7.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-02-28 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Scores on Maslach Burnout Inventory over time | baseline, 4 weeks , 8 weeks
  Survey instruments
Changes in health as measured by scores on the RAND Short-Form 12 over time | baseline, 4 weeks , 8 weeks
  Survey instrument
Changes in fatigue as measured by the Iowa Fatigue Scale over time | baseline, 4 weeks , 8 weeks
  Survey instrument
Changes in mental health symptoms measured by the Depression/Anxiety/Stress Scale (21) over time | baseline, 4 weeks , 8 weeks
  Survey instrument

SECONDARY OUTCOMES:
Change in Serum total antioxidant capacity over time | baseline, 4 weeks, 8 weeks
  Serum laboratory test
Change in Th1 cytokine levels from peripheral blood and culture supernatants over time | baseline, 4 weeks, 8 weeks
  Immunologic tests
Change in Th1 cytokine levels from peripheral blood and culture supernatants | baseline, 4 weeks, 8 weeks
  Immunologic test
Change in Urinary Urolithins over time | baseline, 4 weeks, 8 weeks
  Urinary metabolite of pomegranate
Change in serum total oxidative stress over time | baseline, 4 weeks, 8 weeks
  Serum laboratory test
Change in Th2 cytokine levels from peripheral blood and culture supernatants over time | baseline, 4 weeks, 8 weeks
  Immunologic test
Change in Th17 cytokine levels from peripheral blood and culture supernatants over time | baseline, 4 weeks, 8 weeks
  Immunologic test
Change in TREG cytokine levels from peripheral blood and culture supernatants over time | baseline, 4 weeks, 8 weeks
  Immunologic test

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Mann, MD, MPH, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD.